CLINICAL TRIAL: NCT01175811
Title: A Comparison of Premixed and Basal-Bolus Insulin Intensification Therapies in Patients With Type 2 Diabetes Mellitus With Inadequate Glycaemic Control on Twice-daily Premixed Insulin
Brief Title: A Study Comparing Insulin Intensification Therapies in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13492; F3Z-CR-IOQD (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Metabolic Diseases; Diabetes Mellitus, Type 2; Glargine; Diabetes Mellitus; Insulin LISPRO; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Diseases; Diabetes Mellitus; Insulin Resistance | interventions — insulin lispro, isophane insulin lispro drug combination (25:75); Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Premixed Insulin (Experimental): Twice daily (before breakfast and lunch) insulin lispro mix 50 (50% insulin lispro, 50% insulin lispro protamine suspension [LM50]) and once daily (before dinner) insulin lispro mix 25 (25% insulin lispro, 75% insulin lispro protamine suspension [LM25])
  Interventions: Drug: Insulin Lispro Premix
- Basal-Bolus (Active Comparator): Once daily (bedtime) insulin glargine and three pre-meal insulin lispro
  Interventions: Drug: Insulin Glargine; Drug: Insulin Lispro

INTERVENTIONS:
Drug: Insulin Lispro Premix — Participant dependent dose, administered subcutaneously for 24 weeks
  Other Names: Humalog Mix25; Humalog Mix50; LY275585
  Arms: Premixed Insulin
Drug: Insulin Glargine — Participant dependent dose, administered subcutaneously for 24 weeks
  Arms: Basal-Bolus
Drug: Insulin Lispro — Participant dependent dose, administered subcutaneously for 24 weeks
  Other Names: Humalog; LY275585
  Arms: Basal-Bolus

SUMMARY:
The purpose of the study is to compare the effects on overall glycaemic control of two insulin intensification therapies.

ELIGIBILITY:
Inclusion Criteria:

* Present with type 2 diabetes mellitus
* Have been receiving twice-daily premixed insulin therapy with or without metformin and/or alpha-glucosidase inhibitors, for at least six months prior to study entry
* Have Haemoglobin A1c (HbA1c) >7.0% and <12.0%

Exclusion Criteria:

* Within the last 3 months prior to entry into the study, are taking any non-permitted glucose-lowering agents, or are taking any non-permitted oral antihyperglycaemic medications
* Are pregnant or intend to become pregnant during the course of the study, or are sexually active women of childbearing potential not actively practicing birth control by a method determined by the investigator to be medically acceptable.
* Are women who are breastfeeding.
* Have an irregular sleep/wake cycle (for example, participants who sleep during the day and work during the night).
* Do not regularly consume three meals per day.
* Have a body mass index >35 kilogram per square meter (kg/m^2).
* Have had more than one episode of severe hypoglycaemia within 24 weeks prior to entry into the study.
* Have cardiac disease with a functional status that is Class III or IV
* Have a history of renal or liver disease
* Have used less than or equal to 20 Units per day (U/day) of insulin during the past 90 days for more than 14 days (accumulated).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- China (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kunming
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xi'an
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yeongdeungpo-gu
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuei Shan Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sindian City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yong Kung City

REFERENCES:
- [Derived] Jia W, Xiao X, Ji Q, Ahn KJ, Chuang LM, Bao Y, Pang C, Chen L, Gao F, Tu Y, Li P, Yang J. Comparison of thrice-daily premixed insulin (insulin lispro premix) with basal-bolus (insulin glargine once-daily plus thrice-daily prandial insulin lispro) therapy in east Asian patients with type 2 diabetes insufficiently controlled with twice-daily premixed insulin: an open-label, randomised, controlled trial. Lancet Diabetes Endocrinol. 2015 Apr;3(4):254-62. doi: 10.1016/S2213-8587(15)00041-8. Epub 2015 Mar 6. PMID 25754414

RESULTS

PARTICIPANT FLOW:
Groups:
- Premixed Insulin: Twice daily (breakfast and lunch) insulin lispro mix 50 (LM50) and once daily (dinner) insulin lispro mix 25 (LM25)
  Insulin Lispro Mix: Participant dependent dose, administered subcutaneously for 24 weeks
Period: Overall Study
Arm/Group | Premixed Insulin | Basal-Bolus
Started | 199 | 203
Received at Least 1 Dose of Study Drug | 197 | 202
Completed | 183 | 189
Not Completed | 16 | 14
Not completed — Adverse Event | 1 | 1
Not completed — Entry criteria not met | 3 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Basal-Bolus: Once daily (bedtime) insulin glargine and three pre-meal insulin lispro Insulin Glargine: Participant dependent dose, administered subcutaneously for 24 weeks
  Insulin Lispro: Participant dependent dose, administered subcutaneously for 24 weeks
- Total: Total of all reporting groups
Arm/Group | Premixed Insulin | Basal-Bolus | Total
Number analyzed (Participants) | 199 | 203 | 402
Age Continuous [Mean (Standard Deviation); unit: years] | 59.0 (9.29) | 58.1 (9.05) | 58.6 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 93 | 196
  Male | 96 | 110 | 206
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 199 | 203 | 402
  Non-Asian | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 18 | 20 | 38
  China | 157 | 158 | 315
  Korea, Republic of | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in Haemoglobin A1c (HbA1c) From Baseline to 24 Week Endpoint
Description: Least Squares (LS) means are calculated using mixed model repeating measures (MMRM) with the change from baseline in HbA1c at all post baseline measurement as dependent variables, treatment, country, visit and treatment by visit interaction as fixed effects, baseline HbA1c value as a covariate and participant as a random effect.
Time Frame: Baseline, 24 weeks
Population: Participants in the intent-to-treat population: participants who had been randomized and received at least one dose of study drug and had at least 1 post-baseline evaluable HbA1c data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent HbA1c
Groups:
- Premixed Insulin: Twice daily (before breakfast and lunch) insulin lispro mix 50 (LM50) and once daily (before dinner) insulin lispro mix 25 (LM25)
  Insulin Lispro Mix: Participant dependent dose, administered subcutaneously for 24 weeks
Arm/Group | Premixed Insulin | Basal-Bolus
Number analyzed (Participants) | 197 | 202
percent HbA1c | -1.05 [-1.19 to -0.92] | -1.06 [-1.19 to -0.93]
Statistical Analysis 1: Comparison: Premixed Insulin vs Basal-Bolus; Test type: Superiority or Other; LSmean difference = 0.01, 95% CI 2-sided [-0.14 to 0.16]

2. Secondary Outcome: Change in HbA1c From Baseline to 12 Week Endpoint
Description: as for outcome 1
Time Frame: Baseline, 12 weeks
Population: Participants in the intent-to-treat population: participants who had been randomized and received at least one dose of study drug and who had a baseline and at least 1 post-baseline evaluable HbA1c data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent HbA1c
Arm/Group | Premixed Insulin | Basal-Bolus
Number analyzed (Participants) | 197 | 202
percent HbA1c | -0.96 [-1.10 to -0.82] | -0.96 [-1.10 to -0.82]
Statistical Analysis 1: Comparison: Premixed Insulin vs Basal-Bolus; Test type: Superiority or Other; LSmean Difference = 0.00, 95% CI 2-sided [-0.15 to 0.16]

3. Secondary Outcome: The Percentage of Participants Who Achieved Haemoglobin A1c (HbA1c) Less Than or Equal to 6.5% and Less Than or Equal to 7% at 12 Weeks and 24 Weeks
Description: The Percentage of participants achieving a haemoglobin A1c (HbA1c) less than or equal (<=) to 6.5% or 7% is defined as 100 multiplied by the number of participants with a HbA1c of the cut-off value (6% or 7%) divided by the number of participants exposed to study drug. Participants with missing HbA1c values at endpoint were treated as not achieving the HbA1c goal.
Time Frame: 12 weeks, 24 weeks
Population: Participants in the intent-to-treat population: participants who had been randomized and received at least one dose of study.
Measure: Number; unit: Percentage of participants
Arm/Group | Premixed Insulin | Basal-Bolus
Number analyzed (Participants) | 197 | 202
Percentage of participants
  <=6.5 Percent HbA1c at 12 weeks | 6.1 | 8.9
  <=7.0 Percent HbA1c at 12 weeks | 26.4 | 27.7
  <=6.5 Percent HbA1c at 24 weeks | 9.1 | 11.9
  <=7.0 Percent HbA1c at 24 weeks | 29.9 | 34.2
Statistical Analysis 1: Comparison: Premixed Insulin vs Basal-Bolus; Test type: Superiority or Other; p = 0.344, Fisher Exact — P-value is for the comparison of participants achieving <=6.5% HbA1c at 12 weeks. P-value was not adjusted for multiplicity and should be interpreted as nominal
Statistical Analysis 2: Comparison: Premixed Insulin vs Basal-Bolus; Test type: Superiority or Other; p = 0.822, Fisher Exact — P-value is for the comparison of participants achieving <=7.0% HbA1c at 12 weeks. P-value was not adjusted for multiplicity and should be interpreted as nominal
Statistical Analysis 3: Comparison: Premixed Insulin vs Basal-Bolus; Test type: Superiority or Other; p = 0.417, Fisher Exact — P-value is for the comparison of participants achieving <=6.5% HbA1c at 24 weeks. P-value was not adjusted for multiplicity and should be interpreted as nominal
Statistical Analysis 4: Comparison: Premixed Insulin vs Basal-Bolus; Test type: Superiority or Other; p = 0.392, Fisher Exact — P-value is for the comparison of participants achieving <=7.0% HbA1c at 24 weeks. P-value was not adjusted for multiplicity and should be interpreted as nominal

4. Secondary Outcome: The 7-point Self-monitored Blood Glucose (SMBG) Profiles at Baseline, 12 Weeks and 24 Weeks.
Description: 7-point Self-monitored Blood Glucose (SMBG) Profiles are measures of blood glucose taken 7 times a day at the morning pre-meal, morning 2-hours post-meal, midday pre-meal, midday 2-hours post-meal, evening pre-meal, evening 2-hours post-meal, and 0300 hour [3 am]. Each participant took measures on 3 non-consecutive days and the average was calculated for each of the 7 time points. The mean of the 7-point averages was calculated for all the participants at baseline, Weeks 12 and 24.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Participants in the intent-to-treat population: participants who had been randomized and received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Premixed Insulin | Basal-Bolus
Number analyzed (Participants) | 197 | 202
milligrams per deciliter (mg/dL)
  Morning Pre-meal (Week 0) (n=195, 201) | 155.0 (34.89) | 157.7 (38.81)
  Morning Pre-meal (Week 12) (n=187, 191) | 141.8 (30.78) | 136.5 (31.44)
  Morning Pre-meal (Week 24) (n=177, 186) | 137.4 (24.96) | 132.4 (25.17)
  Morning 2 hours Post-meal (Week 0) (n=194, 201) | 207.1 (54.74) | 213.6 (53.95)
  Morning 2 hours Post-meal (Week 12) (n=187, 190) | 179.6 (46.17) | 176.5 (43.69)
  Morning 2 hours Post-meal (Week 24) (n=176, 184) | 169.7 (39.04) | 165.8 (35.77)
  Midday Pre-meal (Week 0) (n=195, 200) | 160.7 (47.89) | 164.9 (48.71)
  Midday Pre-meal (Week 12) (n=187, 190) | 142.5 (37.27) | 149.4 (41.58)
  Midday Pre-meal (Week 24) (n=177, 186) | 139.5 (31.05) | 142.1 (32.73)
  Midday 2 hours Post-meal (Week 0) (n=194, 201) | 219.7 (54.03) | 227.5 (54.56)
  Midday 2 hours Post-meal (Week 12) (n=186, 189) | 162.5 (41.53) | 177.2 (44.53)
  Midday 2 hours Post-meal (Week 24) (n=175, 184) | 161.9 (38.66) | 171.1 (39.33)
  Evening Pre-meal (Week 0) (n=195, 200) | 186.6 (44.97) | 190.0 (53.41)
  Evening Pre-meal (Week 12) (n=187, 190) | 148.1 (33.74) | 157.6 (42.00)
  Evening Pre-meal (Week 24) (n=177, 186) | 145.0 (30.67) | 151.1 (33.36)
  Evening 2 hours Post-meal (Week 0) (n=194, 201) | 204.8 (54.31) | 209.9 (58.59)
  Evening 2 hours Post-meal (Week 12) (n=186, 190) | 177.1 (45.29) | 176.2 (40.55)
  Evening 2 hours Post-meal (Week 24)(n=176, 185) | 172.0 (38.77) | 165.6 (38.66)
  0300 Hours (3 am) (Week 0) (n=185, 193) | 175.9 (51.97) | 180.0 (54.35)
  0300 Hours (3 am) (Week 12) (n=177, 185) | 150.3 (39.41) | 163.6 (42.42)
  0300 Hours (3 am) (Week 24) (n=171, 179) | 145.1 (31.45) | 155.8 (34.36)

5. Secondary Outcome: Daily Dose of Insulin: Total, Basal, and Prandial
Time Frame: 24 weeks
Population: Participants in the intent-to-treat population: participants who had been randomized and received at least one dose of study drug. Last observation carried forward (LOCF) principle was used.
Measure: Mean (Standard Deviation); unit: International Units (IU)
Arm/Group | Premixed Insulin | Basal-Bolus
Number analyzed (Participants) | 197 | 202
International Units (IU)
  Total Daily Dose | 52.9 (19.72) | 54.0 (19.00)
  Daily Insulin Dose Basal | 31.539 (11.9288) | 24.717 (9.9304)
  Daily Insulin Dose Bolus (prandial) | 21.385 (7.8823) | 29.269 (10.8353)

6. Secondary Outcome: Change in Body Mass Index (BMI) From Baseline to 12 and 24 Weeks
Description: Body mass index is an estimate of body fat based on body weight divided by height squared. Least Squares (LS) means are calculated using mixed model repeating measures (MMRM) using change from baseline in BMI at all post baseline measurement as dependent variables, treatment, country, visit and treatment by visit interaction as fixed effects, baseline BMI value as a covariate and participants as a random effect.
Time Frame: Baseline, 12 weeks, and 24 weeks
Population: Participants in the intent-to-treat population: participants who had been randomized and received at least one dose of study drug and had baseline and at least 1 post-baseline BMI data.
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram per square meter (kg/m^2)
Arm/Group | Premixed Insulin | Basal-Bolus
Number analyzed (Participants) | 197 | 202
kilogram per square meter (kg/m^2)
  Change at 12 weeks | 0.26 [0.16 to 0.37] | 0.20 [0.10 to 0.30]
  Change at 24 weeks | 0.31 [0.19 to 0.42] | 0.29 [0.18 to 0.40]

7. Secondary Outcome: Daily Dose of Insulin Per Kilogram of Body Weight: Total, Basal and Prandial
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: International Units per kilogram (IU/kg)
Arm/Group | Premixed Insulin | Basal-Bolus
Number analyzed (Participants) | 197 | 202
International Units per kilogram (IU/kg)
  Total Daily Dose | 0.738 (0.2477) | 0.760 (0.2694)
  Daily Insulin Dose Basal | 0.440 (0.1498) | 0.348 (0.1390)
  Daily Insulin Dose Bolus (prandial) | 0.298 (0.0994) | 0.412 (0.1542)

8. Secondary Outcome: Percentage of Participants With Hypoglycemic Episodes (Incidence)
Description: Incidence of hypoglycemic episodes is defined as 100 multiplied by the number of participants experiencing a hypoglycemic episode divided by the number of participants exposed to study drug. Hypoglycemic episodes are defined as an event which is associated with reported signs and symptoms of hypoglycemia, and/or a documented blood glucose (BG) concentration of <= 70 mg/dL (3.9 mmol/L).
Time Frame: baseline through 24 weeks
Population: Participants in the safety analyses population: participants who had been randomized and received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Premixed Insulin | Basal-Bolus
Number analyzed (Participants) | 197 | 202
percentage of participants | 54.8 | 55.0

9. Secondary Outcome: The Rate of Hypoglycemic Episodes
Description: The rate of hypoglycemic episodes is defined as the mean number of hypoglycemic episodes per 30 days per participant. Hypoglycemic episodes are defined as an event which is associated with reported signs and symptoms of hypoglycemia, and/or a documented blood glucose (BG) concentration of <= 70 mg/dL (3.9 mmol/L).
Time Frame: baseline through 24 weeks
Population: as for outcome 8
Measure: Mean (Standard Error); unit: hypoglycemic episode/30 days/participant
Arm/Group | Premixed Insulin | Basal-Bolus
Number analyzed (Participants) | 197 | 202
hypoglycemic episode/30 days/participant | 0.468 (1.0417) | 0.409 (0.6668)

10. Secondary Outcome: Percentage of Participants Experiencing a Severe Hypoglycemic Episode
Description: Severe hypoglycemic episode is defined as any event requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. The percentage of participants experiencing a severe hypoglycemic episode is defined as the 100 multiplied by the number of participants experiencing a severe hypoglycemic episode divided by the number of participants exposed to study drug.
Time Frame: baseline through 24 weeks
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Premixed Insulin | Basal-Bolus
Number analyzed (Participants) | 197 | 202
Percentage of participants | 0.0 | 0.0

ADVERSE EVENTS:
Arm/Group | Premixed Insulin | Basal-Bolus
Serious Adverse Events (participants affected / at risk) | 13/197 | 8/202
Other Adverse Events (participants affected / at risk) | 60/197 | 60/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Premixed Insulin (N=197) | Basal-Bolus (N=202)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Premixed Insulin (N=197) | Basal-Bolus (N=202)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 2 (2)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (6)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (6) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 3 (3) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 15 (16) | 17 (19)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (10) | 10 (12)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Weight increased (Investigations) | 3 (3) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (7) | 6 (6)
Headache (Nervous system disorders) | 2 (2) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypogeusia (Nervous system disorders) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days